CLINICAL TRIAL: NCT02897661
Title: Washed Microbiota Transplantation Combining Exclusive Enteral Nutrition Contribute to Nutritional Improvement of Patients With Crohns' Disease
Brief Title: Washed Microbiota Transplantation Improves Nutritional Status of Patients With Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-CN-160814
Record Dates: First submitted 2016-08-14; First posted 2016-09-13 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Crohn's Diseases
Keywords: fecal microbiota transplantation; exclusive enteral nutrition; washed microbiota transplantation; malnutrition
MeSH Terms: conditions — Crohn Disease; Malnutrition

ARMS (2):
- Early WMT and EEN (Experimental): WMT (day1), EEN (day1-15)
  Interventions: Procedure: WMT; Dietary Supplement: EEN
- Late WMT and EEN (Experimental): WMT (day8), EEN (day1-15)
  Interventions: Procedure: WMT; Dietary Supplement: EEN

INTERVENTIONS:
Procedure: WMT — Washed microbiota transplantation (WMT) through mid-gut
Dietary Supplement: EEN — Exclusive enteral nutrition (EEN) through feeding tube

SUMMARY:
Patients with Crohns' disease (CD) are always complicated with malnutrition. Exclusive enteral nutrition (EEN) is an effective treatment to improve nutritional status and induce remission in patients with CD however a reduction in microbiota diversity was the most frequently reported effect of EEN. There was a raised critical question that whether EEN combining microbiota transplantation can bring much more benefits to those CD patients with malnutrition.

Fecal microbiota transplantation (FMT) is an effective way of remodeling microbiota. The improved methodology of FMT in our group since 2014 was different from the traditional manual FMT and was recently coined as washed microbiota transplantation (WMT), which is dependent on the automatic facilities and washing process in a laboratory room with biosafety level 3.

Importantly, the worse nutritional status might decrease the efficacy of FMT. Therefore, there was a raised critical question that when is the proper time to combine WMT for those CD patients requiring EEN. This trial aimed to explore the timing of WMT in CD patients with malnutrition and assess the efficacy and safety of the strategy using WMT combined with EEN in CD patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18 to 65 years with active CD, as defined by Harvey-Bradshaw Index (HBI) score >4;
2. patients accompanied with malnutrition as assessed by Nutritional Risk Screening 2002 (NRS2002) score ≥ 3 or Patient-Generated Subjective Global Assessment (PG-SGA) score ≥ 4;
3. patients with high compliance.

Exclusion Criteria:

1. accompanying with contraindications of enteral nutrition (EN) such as ileus, active gastrointestinal bleeding and shock;
2. severe comorbidities (e.g., Clostridium difficile infection, diabetes, cancer, cardiopulmonary failure and severe liver and kidney diseases;
3. parenteral infection such as urinary infection, pneumonia, etc;
4. steroids or biologicals use within 6 week;
5. intestinal fibrotic stenosis;
6. patients who are pregnant or going to be pregnant;
7. patients with mental disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
changes in hemoglobin | Day 8 and day 15
changes in albumin and prealbumin in g/L | Day 8 and day 15
changes in lymphocyte count in 10^9/L | Day 8 and day 15

SECONDARY OUTCOMES:
rate of clinical remission | day 15
  HBI score ≤ 4

OTHER OUTCOMES:
rate of adverse events | in 1 month following WMT
  abdominal pain, fever, increased frequency of defecation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD; PHD, Study Chair — Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Tjellstrom B, Hogberg L, Stenhammar L, Magnusson KE, Midtvedt T, Norin E, Sundqvist T. Effect of exclusive enteral nutrition on gut microflora function in children with Crohn's disease. Scand J Gastroenterol. 2012 Dec;47(12):1454-9. doi: 10.3109/00365521.2012.703234. Epub 2012 Sep 28. PMID 23016828
- [Background] Cui B, Feng Q, Wang H, Wang M, Peng Z, Li P, Huang G, Liu Z, Wu P, Fan Z, Ji G, Wang X, Wu K, Fan D, Zhang F. Fecal microbiota transplantation through mid-gut for refractory Crohn's disease: safety, feasibility, and efficacy trial results. J Gastroenterol Hepatol. 2015 Jan;30(1):51-8. doi: 10.1111/jgh.12727. PMID 25168749
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Derived] Xiang L, Yu Y, Ding X, Zhang H, Wen Q, Cui B, Zhang F. Exclusive Enteral Nutrition Plus Immediate vs. Delayed Washed Microbiota Transplantation in Crohn's Disease With Malnutrition: A Randomized Pilot Study. Front Med (Lausanne). 2021 Oct 22;8:666062. doi: 10.3389/fmed.2021.666062. eCollection 2021. PMID 34746161